CLINICAL TRIAL: NCT07201103
Title: The Effects of Augmented Reality-Based Exercise Training on Body Awareness, Trunk Appearance Perception, and Exercise Adherence in Adolescents With Idiopathic Scoliosis: A Randomized Controlled Trial
Brief Title: Augmented Reality-Based Exercise Training in Adolescents With Idiopathic Scoliosis
Acronym: AR-SCOLIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Adnan Batuhan Coskun, Asst.Prof.Dr., Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 323S271; TÜBİTAK 1001 Projesi - 323S271 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Adolescent Idiopathic Scoliosis; AR-based Rehabilitation; Augmented Reality Exercise Training; Physiotherapeutic Scoliosis-Specific Exercises (PSSE); Schroth Method; Exercise Adherence; Body Awareness; Trunk Appearance Perception
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated to either the control group (conventional PSSE-Schroth) or the intervention group (AR-assisted PSSE-Schroth). Both groups received supervised exercise training over 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation to reduce assessment bias. Participants and care providers were not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Conventional PSSE-Schroth (Active Comparator): Participants in this group received supervised conventional Physiotherapeutic Scoliosis-Specific Exercises (PSSE-Schroth) for 4 weeks. The program included one 45-minute supervised session per week, complemented by home exercises. Established scoliosis rehabilitation protocols focusing on posture correction, breathing, and spinal alignment were followed.
  Interventions: Behavioral: Conventional PSSE-Schroth
- Experimental - AR-assisted PSSE-Schroth (Experimental): Participants in this group received supervised augmented reality (AR)-assisted Physiotherapeutic Scoliosis-Specific Exercises (PSSE-Schroth) for 4 weeks. The intervention included one 45-minute supervised session per week, supplemented with home exercises. Augmented reality technology was used to provide real-time visual and kinesthetic feedback, aiming to enhance posture correction, breathing patterns, and spinal alignment.
  Interventions: Behavioral: AR-Assisted PSSE-Schroth

INTERVENTIONS:
Behavioral: Conventional PSSE-Schroth — Participants performed conventional Physiotherapeutic Scoliosis-Specific Exercises (PSSE-Schroth) for 4 weeks. The program consisted of one 45-minute supervised session per week complemented by home-based exercises. The exercises focused on posture correction, spinal alignment, and corrective breathing techniques according to standard scoliosis rehabilitation protocols.
  Other Names: Schroth Method
  Arms: Control - Conventional PSSE-Schroth
Behavioral: AR-Assisted PSSE-Schroth — Participants performed Physiotherapeutic Scoliosis-Specific Exercises (PSSE-Schroth) enhanced with augmented reality (AR) support for 4 weeks. The intervention included one 45-minute supervised session per week, plus home-based exercises. The AR system provided real-time visual and kinesthetic feedback during exercise sessions to improve body awareness, trunk appearance perception, and adherence.
  Other Names: Augmented Reality Exercise Training
  Arms: Experimental - AR-assisted PSSE-Schroth

SUMMARY:
This randomized controlled trial investigates the effects of augmented reality (AR)-based exercise training in adolescents with idiopathic scoliosis. Participants are randomly assigned to either a control group receiving conventional Physiotherapeutic Scoliosis-Specific Exercises (PSSE-Schroth) or an intervention group receiving AR-assisted PSSE-Schroth exercises. The primary outcomes include body awareness, trunk appearance perception, and exercise adherence. The study aims to evaluate whether AR-assisted training provides additional benefits over conventional therapy in improving postural control, perception, and compliance in scoliosis management.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional spinal deformity that may negatively affect posture, body image, and adherence to exercise-based rehabilitation. While Physiotherapeutic Scoliosis-Specific Exercises (PSSE-Schroth) are widely accepted as a conservative treatment method, adherence and perception-related factors remain challenging.

This study is designed as a parallel-group, randomized controlled trial comparing conventional PSSE-Schroth exercises with AR-assisted PSSE-Schroth training. A total of 30 adolescents diagnosed with AIS were enrolled and randomized into two groups:

Control Group: received supervised PSSE-Schroth exercises.

Intervention Group: received supervised AR-assisted PSSE-Schroth exercises.

The intervention lasted 12 weeks, and participants were evaluated at baseline and post-intervention.

Primary outcome measures include body awareness (Awareness-Body-Chart), trunk appearance perception (Walter Reed Visual Assessment Scale, Spinal Appearance Questionnaire), and exercise adherence (Exercise Adherence Rating Scale).

Secondary outcome measures include Cobb angle, vertebral rotation, pain intensity, and treatment satisfaction.

The study hypothesizes that AR-assisted PSSE-Schroth training will enhance body awareness, improve trunk appearance perception, and increase adherence compared to conventional methods. This research may provide new insights into integrating digital technologies into scoliosis rehabilitation and contribute to developing innovative, patient-centered approaches in physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

Adolescents clinically diagnosed with idiopathic scoliosis (AIS)

Cobb angle between 10° and 30°

Age range: 10-18 years

No history of spinal surgery

Ability to regularly participate in the exercise program

Signed informed consent obtained from both participants and their parents

Exclusion Criteria:

Diagnosis of neuromuscular, congenital, or secondary scoliosis

Previous history of spinal surgery

Presence of severe cardiovascular, respiratory, or musculoskeletal conditions preventing participation in exercise

Visual, auditory, or perceptual impairments that would hinder participation in augmented reality-based training

Concurrent participation in another physiotherapy or rehabilitation program during the study period

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Awareness (ABC - Vücut Farkındalık Çizelgesi) | Baseline (T0) and 4 weeks after intervention (T4).
  Body awareness will be assessed using the standardized Awareness-Body-Chart (ABC). Participants rate awareness of different body regions, and a total score is calculated. The outcome is the change in total ABC score from baseline (T0) to the end of intervention (T4, 4th week). A higher score indicates greater body awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan B Coşkun, PhD, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, the decision on sharing individual participant data (IPD) is undecided. As the study is supported by TÜBİTAK (The Scientific and Technological Research Council of Turkey), any data sharing must comply with the funder's policies, ethical approval requirements, and national data protection regulations. The research team is committed to transparency and is open to sharing de-identified, anonymized data upon reasonable request from qualified researchers. Such sharing will only take place after publication of the study results, and contingent upon TÜBİTAK's approval and the execution of appropriate data-sharing agreements to ensure participant confidentiality and compliance with legal and ethical standards.

REFERENCES:
- [Background] Yuan W, Shi W, Chen L, Liu D, Lin Y, Li Q, Lu J, Zhang H, Feng Q, Zhang H; Digital Care Study Group. Digital Physiotherapeutic Scoliosis-Specific Exercises for Adolescent Idiopathic Scoliosis: A Randomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2459929. doi: 10.1001/jamanetworkopen.2024.59929. PMID 39964686
- [Background] Cavalcanti, V. C., Ferreira, M. I. d. S., Teichrieb, V., Barioni, R. R., Correia, W. F. M., Da Gama, A. E. F. 2019. "Usability and effects of text, image and audio feedback on exercise correction during augmented reality based motor rehabilitation", Computers & Graphics, 85, 100-10.
- [Background] Kocaman H, Bek N, Kaya MH, Buyukturan B, Yetis M, Buyukturan O. The effectiveness of two different exercise approaches in adolescent idiopathic scoliosis: A single-blind, randomized-controlled trial. PLoS One. 2021 Apr 15;16(4):e0249492. doi: 10.1371/journal.pone.0249492. eCollection 2021. PMID 33857180
- [Background] Buyukturan O, Kaya MH, Alkan H, Buyukturan B, Erbahceci F. Comparison of the efficacy of Schroth and Lyon exercise treatment techniques in adolescent idiopathic scoliosis: A randomized controlled, assessor and statistician blinded study. Musculoskelet Sci Pract. 2024 Aug;72:102952. doi: 10.1016/j.msksp.2024.102952. Epub 2024 Apr 12. PMID 38631273
- [Background] Chen C, Xu J, Li H. Effects of Schroth 3D Exercise on Adolescent Idiopathic Scoliosis: A Systematic Review and Meta-Analysis. Children (Basel). 2024 Jul 1;11(7):806. doi: 10.3390/children11070806. PMID 39062255
- [Background] Schreiber S, Parent EC, Khodayari Moez E, Hedden DM, Hill DL, Moreau M, Lou E, Watkins EM, Southon SC. Schroth Physiotherapeutic Scoliosis-Specific Exercises Added to the Standard of Care Lead to Better Cobb Angle Outcomes in Adolescents with Idiopathic Scoliosis - an Assessor and Statistician Blinded Randomized Controlled Trial. PLoS One. 2016 Dec 29;11(12):e0168746. doi: 10.1371/journal.pone.0168746. eCollection 2016. PMID 28033399
- [Background] Berdishevsky H, Lebel VA, Bettany-Saltikov J, Rigo M, Lebel A, Hennes A, Romano M, Bialek M, M'hango A, Betts T, de Mauroy JC, Durmala J. Physiotherapy scoliosis-specific exercises - a comprehensive review of seven major schools. Scoliosis Spinal Disord. 2016 Aug 4;11:20. doi: 10.1186/s13013-016-0076-9. eCollection 2016. PMID 27525315